CLINICAL TRIAL: NCT01231477
Title: Effects of Inhalation Anaesthesia With Sevoflurane on Cytokine Response in Patients Submitted to Otorhinolaryngological Surgery
Brief Title: Cytokines and Sevoflurane During Surgery
Status: Completed | Type: Observational
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Other Study IDs: JEO4531
Record Dates: First submitted 2010-10-29; First posted 2010-11-01 (Estimated); Last update posted 2010-11-01 (Estimated); Status verified 2010-10

CONDITIONS: Cytokines; Inflammatory; Sevoflurane
Keywords: anaesthetic techniques, inhalation; sevoflurane; Cytokines; Immune response
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Volunteers: Healthy volunteers not submitted to anesthesia nor surgery.
- Sevoflurane Group: This group was submitted to inhalational anesthesia with sevoflurane and otorhinolaryngological surgery.

SUMMARY:
The aim of the present study was to evaluate the effects of anaesthesia with sevoflurane and surgery on cytokines response.

ELIGIBILITY:
Inclusion Criteria:

* both gender, ASA I physical status, 18-50 years old, tympanoplasty and septoplasty.

Exclusion Criteria:

* Malignant or genetical diseases; diabetes; smoking; elicit drugs, recent RX radiation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Thirty adult patients ASA I physical status were allocated in 2 grups: 15 volunteers, not submitted to anesthesia and surgery, and 15 patients scheduled for tympanoplasty or septoplasty anesthetized with sevoflurane at 2,5%. Blood samples were drawn at 4 moments: before induction of anaesthesia, before surgery, at 120 minutes after anaesthesia induction, and on the postoperative first day. Blood samples from volunteers were drawn only once.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose EB Orosz, MD, Principal Investigator — Botucatu Medical School
Locations (1):
- Botucatu Medical School, Botucatu, São Paulo, Brazil